CLINICAL TRIAL: NCT01705873
Title: Retrospective Analysis on the Risk of Cardiovascular (CV) Events in HIV- Infected Subjects From Latin America Treated With a Lopinavir/Ritonavir (LPV/r) Based HAART Regimen vs. an Efavirenz (EFV) Based HAART Regimen
Brief Title: Analysis on the Risk of Cardiovascular Events in HIV- Infected Subjects Treated With LPV/r Based HAART Regimen vs. an EFV Based Regimen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helios Salud (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Isabel Cassetti, MD, Helios Salud
Other Study IDs: ANV-10-0165
Record Dates: First submitted 2012-10-05; First posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: HIV; Hypercholesterolemia; Dyslipidemia
Keywords: HIV; cardiovascular; risk; mortality
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LPV/r: LPV/r based HAART
- Efavirenz: EFV first line based HAART

SUMMARY:
The objective of this study is to evaluate changes in Framingham score (from low to moderate, from moderate to high) based on changes in lipid profile and other parameters from baseline to 48 weeks of HAART in naïve patients or patients in second line of treatment, considering LPV/r vs EFV based HAART. The null hyphotesis is that there is an increased Framingham score in patients treated with LPV/r as second line treatment and in patients treated with LPV/r or EFV regimen as first line treatments.

DETAILED DESCRIPTION:
Study design and duration: Retrospective comparative study. Estimated time of enrollment: 12 months.

Procedure: Retrospective review of clinical charts: LPV/r (n = 100) and EFV (a randomly selected representative sample of patients under EFV treatment: 200 patients approximately.). Each patient can only be included in one arm of the study (cannot switch EFV to LPV/r or from LPV/r to EFV)

Subject population

LPV/r (n = 100) and EFV (a randomly selected representative sample of patients under EFV treatment: 200 patients approximately.). Each patient can only be included in one arm of the study (cannot switch EFV to LPV/r or from LPV/r to EFV)

Study Objectives:

Primary Objectives

1)Changes in Framingham score (from low to moderate, from moderate to high) based on changes in lipid profile and other parameters from baseline to 48 weeks of HAART in naïve patients or patients in second line of treatment Secondary Objectives

1. Risk assessment hazard of CV events in HIV- infected subjects treated with a LPV/r as second line and EFV and LPV/r first line based HAART regimen in the whole population under study and in the female and male subpopulations.
2. Assessment for 10- year risk of developing hard cardiovascular events (myocardial infarction and coronary death) in HIV- infected subjects treated with a LPV/r ( 1° o 2° line) and EFV first line based HAART regimen
3. Overall mortality (including CV events) in HIV- infected subjects treated with a LPV/r as second line and EFV and LPV/r first line based HAART regimen
4. Evolution of lipid profile (total cholesterol, HDL, LDL and triglicerides) and lipid lowering agents requirement: baseline vs. 48 weeks after the initiation of a LPV/r second line based HAART regimen and those on an LPV/r and EFV first line based HAART regimen
5. Assesment of CD4 T-cell count and viral load at baseline and at 48 weeks in each regimen.

ELIGIBILITY:
Inclusion criteria

1. HIV positive patients (confirmation with ELISA + W. blot required).
2. Age ≥ 18 years.
3. Naïve or experienced with antiretroviral drugs.
4. LPV/r or EFV as first line regimen.
5. In patients with a LPV/r second line HAART regimen, prior exposure to any NNRTI regimen is acceptable.
6. Time of exposure to LPV/r or EFV of at least 48 weeks.

Exclusion criteria:

1. Age < 18 yrs.
2. Already LPV/r treatment at admission in our institution (that prevents assessment of baseline lipid profile and CV risk when patient receives the "first dose" of either LPV/r )
3. Patients that had received LPV/r only during they pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients with first line HAART with EFV or LPV/r or second line HAART with LPV/r
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Risk for CV events | Per year
  Changes in Framingham risk for CV events (from low to moderate, from moderate to high) based on changes in lipid parameters from baseline at 6, 12, Q12 months after the initiation of a LPV/r based HAART regimen in the whole population under study.Participants will be followed for an average of 24 months .
Risk for CV events | Per year
  Changes in Framingham risk for CV events (from low to moderate, from moderate to high) based on changes in lipid parameters from baseline at 6, 12, Q12 months after the initiation of a LPV/r based HAART regimen in male subpopulation.Participants will be followed for an average of 24 months .
Risk for CV events | Per year
  Changes in Framingham risk for CV events (from low to moderate, from moderate to high) based on changes in lipid parameters from baseline at 6, 12, Q12 months after the initiation of a LPV/r based HAART regimen in female subpopulation. Participants will be followed for an average of 24 months .

SECONDARY OUTCOMES:
All cause mortality | Per year
  Overall mortality (including CV events) in HIV- infected subjects treated with a LPV/r as second line and EFV and LPV/r first line based HAART regimen in the whole population under study. Participants will be followed for an average of 24 months .
All cause mortality | Per year
  Overall mortality (including CV events) in HIV- infected subjects treated with a LPV/r as second line and EFV and LPV/r first line based HAART regimen in male subpopulation.Participants will be followed for an average of 24 months .
All cause mortality | Per year
  Overall mortality (including CV events) in HIV- infected subjects treated with a LPV/r as second line and EFV and LPV/r first line based HAART regimen in female subpopulation. Participants will be followed for an average of 24 months .

OTHER OUTCOMES:
Evolution of lipid profile | Per year
  Evolution of lipid profile (total cholesterol, HDL, LDL and triglicerides) and lipid lowering agents requirement from baseline at 6, 12, Q12 months after the initiation of a LPV/r second line based HAART regimen and those on an LPV/r or EFV first line based HAART regimen in the whole population under study. Participants will be followed for an average of 24 months .
Evolution of lipid profile | Per year
  Evolution of lipid profile (total cholesterol, HDL, LDL and triglicerides) and lipid lowering agents requirement from baseline at 6, 12, Q12 months after the initiation of a LPV/r second line based HAART regimen and those on an LPV/r or EFV first line based HAART regimen in male subpopulation. Participants will be followed for an average of 24 months .
Evolution of lipid profile | Per year
  Evolution of lipid profile (total cholesterol, HDL, LDL and triglicerides) and lipid lowering agents requirement from baseline at 6, 12, Q12 months after the initiation of a LPV/r second line based HAART regimen and those on an LPV/r or EFV first line based HAART regimen in female subpopulation. Participants will be followed for an average of 24 months .

CONTACTS AND LOCATIONS:
Overall Officials: Lidia I Cassetti, MD, Principal Investigator — Helios Salud; Diego M Cecchini, PhD, Study Chair — Helios Salud
Locations (1):
- Helios Salud, Buenos Aires, Argentina

REFERENCES:
- [Derived] Cecchini D, Mattioli MI, Cassetti J, Chan D, Cassetti I. Evolution of Framingham cardiovascular risk score in HIV-infected patients initiating EFV- and LPV/r-based HAART in a Latin American cohort. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19547. doi: 10.7448/IAS.17.4.19547. eCollection 2014. PMID 25394054